CLINICAL TRIAL: NCT01429181
Title: Pilot Study to Evaluate Efficacy, Tolerability and Safety Nonracemic Methadone HCl in Patients With Chronic Peripheral Neuropathic Pain: Double-Blind, Placebo-Controlled, Crossover Study Followed by Open-Label, Single-Arm Extension
Brief Title: Efficacy & Safety Study of Nonracemic Methadone for the Relief of Chronic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MetaPharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP10-001
Record Dates: First submitted 2011-08-31; First posted 2011-09-05 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non Racemic Methadone (Experimental): Non-Racemic Methadone Hydrochloride 5 mg Capsules containing a non-racemic mixture of methadone isomers.
  Interventions: Drug: Non-racemic mixture of methadone HCl
- Placebo (Placebo Comparator): Matching placebo capsules
  Interventions: Drug: Non-racemic mixture of methadone HCl

INTERVENTIONS:
Drug: Non-racemic mixture of methadone HCl — Non-racemic mixture of methadone HCl capsules, 5 mg

SUMMARY:
There is a growing evidence that the d-isomer of methadone is effective in treating neuropathic pain while the l-isomer of methadone is the only effective isomer of methadone for treating somatic pain. This study will examine a combination of different amounts of the d- and l-isomers of methadone specifically tailored to the chronic peripheral neuropathic pain. Non-racemic mixture of methadone isomers will be tested in this pilot efficacy and safety study.

This study will evaluate effect of the three doses of the non-racemic mixture of methadone hydrochloride patients with chronic peripheral neuropathic pain compared with a placebo. The study will also examine the minimally effective and maximally tolerated doses of the non-racemic mixture of methadone. Finally, the safety and tolerability of the non-racemic methadone therapy will be evaluated.

DETAILED DESCRIPTION:
Objectives:

* To evaluate effect of the three doses of the non-racemic methadone HCl on the metrics of pain intensity in comparison to placebo.
* To determine minimally effective and maximally tolerated doses of non-racemic methadone HCl for the treatment of diabetic peripheral neuropathic pain.
* To evaluate safety and tolerability of non-racemic methadone HCl therapy.

Study Design:

This is a pilot efficacy and safety study comprised of two parts.

Part I is a double-blind, placebo-controlled, crossover study of three daily doses (15 mg, 30 mg and 40 mg) of non-racemic methadone compared with placebo. Two lower doses (15 mg and 30 mg) will be administered for 1 week. The final dose (40 mg) will be administered for 2 weeks. After receiving three consecutive doses of the assigned drug the subjects will be switched to another regimen. Two 28-day treatment periods will be separated by a 14-day washout (drug-free) interval.

Subjects will be randomly assigned to one of the two treatment sequences:

Sequence 1: non-racemic methadone HCl (Period 1) followed by Placebo (Period 2); Sequence 2: Placebo (Period 1) followed by non-racemic methadone HCl (Period 2).

Subjects completing Part I will be enrolled into the open-label, single-arm extension. Subjects discontinuing the study while on placebo may also be eligible for the enrollment. During the 6-week extension phase (Part II of the study) subjects will be treated with non-racemic methadone HCl with continuous dose titration driven by the clinical response (degree of pain relief) and reported adverse events. The Parts I and II will be separated by a 14-day washout (study drug-free) interval.

Number of Patients:

Up to fifty (50) subjects diagnosed with neuropathic pain associated with diabetic peripheral neuropathy will be enrolled in the study; approximately 30 subjects are expected to complete Study Part I. Enrollment will be terminated when this completion target is achieved.

Study Duration:

The duration of Study Part I is approximately 12 weeks, the duration of Study Part II is approximately 6 weeks. A total study duration (including screening and final evaluations) is expected to be approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older;
* Female with a negative serum βhCG pregnancy test
* Female of non-childbearing potential (postmenopausal or surgically sterile) OR female of child-bearing potential agreed to use the protocol-approved contraceptive method
* Documented diagnosis of neuropathic pain associated with diabetic peripheral neuropathy for at least 6 months
* Average daily pain severity score >=4 for the seven days prior to randomization (based on an 11-point numerical rating scale where 0= no pain and 10=worst possible pain)
* Score >= 40 mm on the VAS of the Short Form McGill Pain Questionnaire (SF-MPQ) at screening and randomization visits
* Stable doses (for at least three weeks) of non-opioid analgesics including NSAIDS, corticosteroids, gabapentin, pregabalin or antidepressants prescribed for the purposes of pain control or pain treatment naïve
* Willing to refrain from any pain-relieving drugs other than the protocol-approved rescue medications (acetaminophen, <= 3 g daily or aspirin <= 325 mg daily) during the screening phase and the course of the study
* Willing to limit alcohol consumption during the study according to protocol requirements
* Able to understand and complete study diary and questionnaires
* Willing to give informed consent prior to entry into the study

Exclusion Criteria:

* A documented neuropathy of any cause other than diabetic peripheral neuropathy
* A severe intermittent pain for reasons other than radiculopathy (e.g., migraine attacks)
* History of head injury and/or increased intracranial pressure
* Any neurologic disorder unrelated to diabetic peripheral neuropathy
* Non-adequate renal and/or hepatic function as follows: Serum creatinine > 1.5 x ULN (upper limit of normal range) Liver enzymes (ALT and AST) > 2 x ULN
* Any other know laboratory abnormality that, in the investigator's opinion, would contraindicate study participation
* Chronic hepatitis B, hepatitis C, or HIV infection
* Abnormal cognition defined as obvious clinical findings of state of arousal, confusion and memory or concentration deficit.
* Recent history (within the previous 12 months) of respiratory depression, acute bronchial asthma or hypercarbia, or any other severe pulmonary or respiratory disease
* Recent history (within the previous 12 months) of sleep apnea
* Any hemostatic disorders or a current treatment with anticoagulants;
* Unstable cardiovascular disease or symptomatic peripheral vascular disease
* Hypotension: sitting or standing systolic blood pressure <= 90 mmHg and/or diastolic blood pressure <= 60 mmHg at screening and/or orthostatic hypotension (defined as a difference between sitting and standing systolic blood pressure >20 mmHg and/or a difference between sitting and standing diastolic blood pressure >10 mmHg)
* Any clinically important ECG abnormality (including QT interval exceeding 450 ms)
* Recent history (within the last 12 months) of risk factors for development of prolonged QT interval, including cardiac hypertrophy, concomitant diuretic use, hypocalcemia, hypomagnesemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in average daily pain scores | From Baseline to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Mironer, MD, Study Director — MetaPharm, Inc.